CLINICAL TRIAL: NCT07350837
Title: An Early-Phase Study of AZD0120 (Also Known as GC012F), a Chimeric Antigen Receptor-T Cell (CAR-T) Therapy Targeting CD19 and B Cell Maturation Antigen (BCMA), for Desensitization in Highly Sensitized Participants With End Stage Kidney Disease Awaiting Kidney Transplant
Brief Title: CAR-T Therapy Targeting CD19 and BCMA in Highly Sensitized Kidney Transplant Participants
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Gang Chen, Ph.D, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D831FFS0001
Record Dates: First submitted 2025-12-29; First posted 2026-01-20 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-12

CONDITIONS: Highly Sensitized Patients Awaiting Kidney Transplant
Keywords: Investigator-Initiated Trial; End-stage kidney disease; Dual directed CD19/BCMA CAR-T desensitization therapy; Kidney Transplantation
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: In this study, a single dose group is planned for the CAR-T cell infusion dose, and this study will enroll up to approximately 12 participants into 2 cohorts: approximately 6 highly sensitized participants with living donors (Cohort 1) and approximately 6 highly sensitized participants without living donors (Cohort 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZD0120 CAR-T Cell Injection (Experimental): This study is An Early Exploratory. The main purpose is an IIT clinical trial to evaluate the safety, tolerability, and efficacy of AZD0120 in highly sensitized adult participants with ESKD awaiting kidney transplant.
  Interventions: Drug: AZD0120

INTERVENTIONS:
Drug: AZD0120 — Treatment duration: A single dose of AZD0120 via IV infusion

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and efficacy of AZD0120 in highly sensitized adult participants with ESKD awaiting kidney transplant-who, as assessed by investigators, are improbable desensitization through conventional treatments (e.g., plasmapheresis and immunoadsorption)- with or without living donors.

DETAILED DESCRIPTION:
This is a single-arm, open-label, early-phase clinical study of AZD0120, a dual-directed CD19/BCMA CAR-T therapy in highly sensitized adult participants with ESKD awaiting kidney transplant. This study aims to evaluate the safety, tolerability, and efficacy of AZD0120 in highly sensitized adult participants with end-stage kidney disease (ESKD) awaiting kidney transplantation-who, as assessed by investigators, are improbable desensitization through conventional treatments (e.g., plasmapheresis and immunoadsorption)-with the participants divided into Cohort 1 (with living donors) and Cohort 2 (without living donors).

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult men or women aged 18 to 65 years with end-stage kidney disease who are waiting for kidney transplant and require desensitization to enable safe kidney transplant.

  2. Cohort 1:
* A living donor who meets criteria for kidney donation based on national and local center-specific guidelines has been identified
* Highly sensitized participants with a requirement of positive flow cytometry crossmatch, resulting from at least one DSA detected using Luminex SAB during or before Screening
* A positive virtual crossmatch, using Luminex SAB (MFI ≥ 2000), obtained within 30 days of Screening and during Screening

Cohort 2:

* PRA greater than or equal to 80% which is consistent with highly sensitized based on national criteria
* At least one anti-HLA antibody that is unacceptable for kidney transplantation 3. High-resolution HLA typing for both the recipient and the donor within 2 years of Screening.

  4. The participant is currently eligible for transplantation according to local standards if a graft becomes available upon completion of treatment with the study intervention.

  5. Hemoglobin ≥ 8 g/dL. 6. ANC ≥ 800/μL. 7. Absolute lymphocyte count ≥ 2000/μL or CD3 T cell count ≥ 500/μL. 8. Platelet count ≥ 75000/μL. 9. Vaccinations must be up to date in accordance with the national and local center guidance for transplant participants.

  10. Positive for EBV capsid IgG. 11. Testing for latent TB infection must be negative within 3 months prior to Screening. Testing should be conducted using either a purified protein derivative or an IFN-γ release assay (ie, QuantiFERON-TB or T-SPOT.TB). Participants with a positive test for latent TB infection must complete appropriate therapy for LTBI.

A participant is considered eligible if he/she has a negative test for LTBI within 3 months prior to Screening, or if he/she has completed appropriate LTBI therapy prior to transplantation. Treatment for latent TB infection should follow national guidelines.

12. Participants must be willing to be hospitalized for at least 2 weeks from the time of AZD0120 infusion and must reside within 2 hours of the hospital for an additional 2 weeks following hospital discharge.

13. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

14. Contraceptive use by male and female participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

15. Nonsterilized male participants who are sexually active with female partner of childbearing potential (See Appendix D for details):

(a)Must agree to use one highly effective method of birth control for at least 3 years post AZD0120 infusion.

(b)For participants who receive LDC but not AZD0120, the contraception time lasts from enrollment until 6 months after the last dose of LDC.

(c)Must refrain from fathering a child or donating sperm within 3 years post AZD0120 infusion.

(d)Female partner of a male participant must use one highly effective method of birth control for at least 3 years post AZD0120 infusion.

16. Female participants (See Appendix D for details):

1. FOCBP who are sexually active with a non-sterilized male partner must agree to use one highly effective method of birth control for at least 3 years post AZD0120 infusion. For FOCBP participants who receive LDC but not AZD0120, the contraception time lasts from enrollment until 12 months after the last dose of LDC. Cessation of contraception after this point should be discussed with a responsible physician.
2. All FOCBP must have a negative serum pregnancy test result 3 days prior to enrollment at Screening.
3. Must refrain from donating ova within 3 years post AZD0120 infusion.

   Exclusion Criteria:
   * 1. Previous solid organ (except kidney) or bone marrow transplant. 2. Complement 3 glomerulopathy, immune-complex mediated membranoproliferative glomerulonephritis, or focal and segmental glomerulosclerosis as the cause of ESKD in the native kidney.

     3. Severe peripheral arterial disease is defined by the presence of resting pain and/or non healing skin ulcers.

     4. History of recurrent UTI; 2 in 6 months or 3 in one year. 5. Active invasive bacterial, viral or fungal infection. Additionally, any infection requiring hospitalization and IV antibiotics within 4 weeks of Screening or PO antibiotics within 2 weeks.

     6. History of HIV regardless of treatment. 7. Evidence of active hepatitis B infection based on positive HBsAg or positive core antibody (anti HBc): participants with positive anti-HBc but negative HBsAg may be enrolled if the HBV DNA test result is negative during the Screening Period.

     8. Evidence of active hepatitis C infection - Positive HCV antibody: Participants with positive HCV antibody and negative HCV RNA test during the Screening Period and absence of cirrhosis may be enrolled.

     9. Detectable viral load for CMV, EBV, BKV or SARS-CoV-2, as determined by PCR. 10. CMV serology incompatible with donor (eg, a recipient with a CMV negative serology should not receive an organ from a CMV positive donor).

     11. History of cirrhosis or severe liver disease, including abnormal liver profile (AST, ALT, or total bilirubin > 3 × ULN at Screening, except for participants whose hyperbilirubinemia is attributed to Gilbert's syndrome).

     12. History of sickle cell disease or systemic amyloidosis. 13. Any chronic illness requiring uninterrupted anticoagulation or antiplatelet therapy, except for clinical stable and asymptomatic conditions (eg, chronic atrial fibrillation).

     14. Active and severe disease requiring prolonged immunosuppressive therapy, except for low dose glucocorticoids (prednisone or prednisone equivalent < 10 mg/day).

     15. Receiving ongoing immunosuppressive treatment, including corticosteroids (excepting < 10 mg/d of prednisone or prednisone equivalent), IV immunoglobulin, CYC, mycophenolic acid, or azathioprine, from 90 days prior to Screening.

     16. CNI use within 14 days prior to Screening. 17. Any B cell depleting or monoclonal antibody therapy within 6 months prior to enrollment.

     18. Cardiac clearance for transplant > 6 months old and/or any of the following conditions: NYHA Class III or IV heart failure, unstable angina, LVEF < 40%, a history of recent (within 6 months of Screening) myocardial infarction or presence of implantable cardioverter/defibrillators and/or biventricular pacing.

     19. Moderate-severe pulmonary function abnormality, defined as resting oxygen saturation < 92% on room air or FEV1, total lung capacity, or DLCO (after correction for hemoglobin) < 50% of predicted values within 6 months of Screening.

     20. Known life-threatening allergies, hypersensitivity, or intolerance to AZD0120 or its excipients, including DMSO.

     21. Pregnant, breastfeeding, or planning to become pregnant while enrolled in this study or within 3 years after receiving study intervention.

     22. Plans to father a child while enrolled in this study or within 3 years after receiving study intervention.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of treatment-related adverse events AE/SAE | Through study completion, an average of 3 years
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.A SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria listed:Results in death and life-threatening.
Occurrence of DLTs. | Through study completion, an average of 3 years
  Dose toxicity is defined as any TEAE that meets the following criteria which cannot be attributed to the disease under study. Dose toxicity will be evaluated according to the ASTCT criteria, and the NCI CTCAE Version 5.0.

SECONDARY OUTCOMES:
Assessment of CAR transgene levels of AZD0120 in peripheral blood over time by ddPCR. | Through study completion, an average of 3 years
  CK CAR transgene levels by ddPCR
Maximum plasma concentration (Cmax) | Through study completion, an average of 3 years
  Cytokinetics (CK) profile of AZD0120 CAR-T celltherapy
Time to maximum plasma concentration (Tmax) | Through study completion, an average of 3 years
  Cytokinetics (CK) profile of AZD0120 CAR-T celltherapy
Last detectable time point（AUC0-28d） | Through study completion, an average of 3 years
  Cytokinetics (CK) profile of AZD0120 CAR-T celltherapy
Last detectable time point（Tlast） | Through study completion, an average of 3 years
  Cytokinetics (CK) profile of AZD0120 CAR-T celltherapy
Last quantifiable concentratione (Clast) | Through study completion, an average of 3 years
  Cytokinetics (CK) profile of AZD0120 CAR-T celltherapy
Circulating soluble BCMA protein levels | Through study completion, an average of 3 years
  Blood will be collected for the measurement of the pharmacodynamics parameters
Depletion of BCMA-expressing B cells | Through study completion, an average of 3 years
  Blood will be collected for the measurement of the pharmacodynamics parameters
Depletion of CD19-expressing B cells | Through study completion, an average of 3 years
  Blood will be collected for the measurement of the pharmacodynamics parameters
Lymphocyte subsets | Through study completion, an average of 3 years
  To evaluate immune cell and signaling responses in peripheral blood after AZD0120 infusion
Time to recovery of lymphocytes and B cells to baseline | Through study completion, an average of 3 years
  To evaluate immune cell and signaling responses in peripheral blood after AZD0120 infusion
Levels of cytokine in peripheral blood IL1, IL2, IL4, IL6, IL8, IL10, IL12, IL13, IFN-γ, and TNF-α | Through study completion, an average of 3 years
  To evaluate immune cell and signaling responses in peripheral blood after AZD0120 infusion
Change from baseline in serum immunoglobulin concentration (including IgG, IgM, IgA, and IgE and IgG subclasses 1-4) | Through study completion, an average of 3 years
  To evaluate immune cell and signaling responses in peripheral blood after AZD0120 infusion
Time to nadir and recovery of IgG | Through study completion, an average of 3 years
  To evaluate immune cell and signaling responses in peripheral blood after AZD0120 infusion
Change from baseline in vaccination titers for MMR(measles, mumps, and rubella (vaccine)) | Through study completion, an average of 3 years
  To measure pharmacodynamics parameters
Change from baseline in vaccination titers for VZV(varicellazoster virus) | Through study completion, an average of 3 years
  To measure pharmacodynamics parameters
Change from baseline in vaccination titers for Tetanus | Through study completion, an average of 3 years
  To measure pharmacodynamics parameters
Change from baseline in vaccination titers for HBV | Through study completion, an average of 3 years
  To measure pharmacodynamics parameters
Flow cytometry for CD19 (pan B cell marker), CD20 (pan B cell marker), CD138 (plasma cells), CD23 (follicular dendritic cells), CD3 (T cells), BCMA (plasma cells), and CD68 (macrophages) | Through study completion, an average of 3 years
  To evaluate cell composition in the lymphatic tissues after AZD01210 infusion in participants who receive kidney transplant.
The incidence of anti CAR AZD0120 antibody response through the duration of the study | Through study completion, an average of 3 years
  To evaluate immunogenicity of AZD0120
The incidence of anti CAR AZD0120 antibody titer through the duration of the study | Through study completion, an average of 3 years
  To evaluate immunogenicity of AZD0120
The incidence of anti CAR AZD0120 antibody category of response through the duration of the study | Through study completion, an average of 3 years
  To evaluate immunogenicity of AZD0120
Proportion of participants who achieve a negative virtual crossmatch based on anti-HLA antibodies Luminex assay | Through study completion, an average of 3 years
  To evaluate the clinical efficacy of AZD0120 in reducing DSA and improving HLA compatibility
Proportion of participants who achieve a negative flow cytometry crossmatch | Through study completion, an average of 3 years
  To evaluate the clinical efficacy of AZD0120 in reducing DSA and improving HLA compatibility
Proportion of participants who achieve a negative CDC crossmatch | Through study completion, an average of 3 years
  To evaluate the clinical efficacy of AZD0120 in reducing DSA and improving HLA compatibility
Percentage and absolute decrease in MFI of Class I and II anti HLA antibodies from baseline to transplantation or the end of follow-up | Through study completion, an average of 3 years
  To evaluate the clinical efficacy of AZD0120 in reducing DSA and improving HLA compatibility
Decline in MFI of Class I and II anti HLA antibodies to MFI < 2000, < 3000, < 5000. | Through study completion, an average of 3 years
  To evaluate the clinical efficacy of AZD0120 in reducing DSA and improving HLA compatibility
Number and proportion of anti HLA antibodies unacceptable for kidney transplantation that were removed. | Through study completion, an average of 3 years
  To evaluate the clinical efficacy of AZD0120 in reducing DSA and improving HLA compatibility
Number and proportion of DSAs removed | Through study completion, an average of 3 years
  To evaluate the clinical efficacy of AZD0120 in reducing DSA and improving HLA compatibility
Proportion of participants achieving ≥ doubling of donor availability based on national PRA. | Through study completion, an average of 3 years
  To evaluate the clinical efficacy of AZD0120 in reducing DSA and improving HLA compatibility
Change in national PRA from baseline over time until kidney transplantation or the end of follow-up, with and without serial dilutions. | Through study completion, an average of 3 years
  To evaluate the clinical efficacy of AZD0120 in reducing DSA and improving HLA compatibility
Time to anti-HLA antibody nadir. | Through study completion, an average of 3 years
  To evaluate the clinical efficacy of AZD0120 in reducing DSA and improving HLA compatibility

CONTACTS AND LOCATIONS:
Overall Officials: Gang Chen, Principal Investigator — Tongji Hospital, Tongji Medical Collage of Huazhong University of Science & Technology
Locations (1):
- Tongji Hospital, Tongji Medical Collage of Huazhong University of Science & Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No